CLINICAL TRIAL: NCT06987890
Title: Practical Geriatric Assessment in Older Adults With Non-Small Cell Lung Cancer Undergoing Stereotactic Body Radiation Therapy
Acronym: Lung-GAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond Mak, Associate Professor of Radiation Oncology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-009
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer (NSCLC); Geriatric Assessment; Stereotactic Body Radiation Therapy (SBRT)
Keywords: Lung Cancer; Geriatric
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Prostaglandins A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGA IMPLEMENTED IN NSCLC WITH SBRT (Experimental): Providers will be made aware of PGA results and all recommended referrals based on PGA results. Providers will be reminded weekly for up to one month regarding these recommendations.
  Interventions: Other: Practical Geriatric Assessment
- SUPPORTIVE CARE WITHOUT PGA IN NSCLC WITH SBRT (No Intervention): Though PGA questions will be completed to characterize baseline impairment, providers will not be notified of PGA results or recommended referrals based on PGA results. Providers will assess for geriatric impairment at their discretion, and will make any service referrals they deem necessary, also at their discretion.

INTERVENTIONS:
Other: Practical Geriatric Assessment — The Practical Geriatric Assessment (PGA) is an abridged version of the Comprehensive Geriatric Assessment (CGA). This tool can be completed by any provider within 10-25 minutes while still capturing the key domains of the CGA. This screening tool, which is now recommended by American Society of Clinical Oncology (ASCO), the International Society for Geriatric Oncology (SIOG), and the Cancer & Aging Research Group (CARG), has the potential capacity to delineate relevant baseline features in geriatric populations without creating undue provider burden.
  Other Names: PGA
  Arms: PGA IMPLEMENTED IN NSCLC WITH SBRT

SUMMARY:
National guidelines recommend that older adults with cancer undergo a special health assessment before starting cancer treatment. This type of assessment evaluates physical function, nutrition, social support, psychological well-being, medical conditions (both cancer-related and non-cancer-related), and cognitive function. The results can help doctors make better treatment decisions and determine whether additional support services-such as nutrition counseling, physical therapy, or social work-would be beneficial. Even though these assessments are recommended, they are not typically used because they need to be performed by a specialist and can take over an hour to complete. Given these challenges, a 10-15-minute assessment called the Practical Geriatric Assessment (PGA) was recently developed. The PGA can be completed by any healthcare provider and helps identify older adults who may need extra support alongside their cancer treatment. While the PGA has the potential to make geriatric assessments more accessible, the investigators do not yet know whether patients will find it useful or easy to complete.

Additionally, it is unclear whether using the PGA will lead to more referrals for recommended supportive care services. This study aims to address these questions. The investigators will evaluate whether using the PGA impacts the number of patients referred to recommended supportive care services. Investigators will also evaluate how participants feel about completing the PGA, including how easy or difficult it is, and to assess the feasibility of implementing this survey on a larger scale. Finally, the investigators will use facial photographs and audio-visual data from the PGA to develop and evaluate artificial intelligence algorithm(s) to identify vulnerable patients who might benefit from additional supportive care services.

DETAILED DESCRIPTION:
Comprehensive geriatric assessment (CGA) is one proven mechanism for delineating baseline care needs and improving outcomes in older adults with lung cancer. This type of geriatrician-led assessment, which captures functional ability, health, and socio-environmental situation, can be used to identify vulnerable older adults for whom tailored interventions might optimize care. However, CGA can be resource-intensive to perform, and may not practically possible in all settings, particularly given national shortages in geriatricians. At BWH/DFCI, retrospective work among patients with stage I-II NSCLC suggests fewer than 5% of patients receive CGA, despite 76% meeting national guidelines for this type of evaluation. These findings underscore the practical challenges of assessing geriatric needs, even in high-resource settings.

To address these barriers, abridged instruments capturing the key domains of the CGA which can be completed by any provider within 10-25 minutes have recently been developed, including the practical geriatric assessment (PGA) tool. This screening tool, which is now recommended by American Society of Clinical Oncology (ASCO), the International Society for Geriatric Oncology (SIOG), and the Cancer & Aging Research Group (CARG), has the potential capacity to delineate relevant baseline features in geriatric populations without creating undue provider burden. However, the feasibility of implementing the PGA and its acceptability to patients remain unclear. Further, relationships between the PGA and salient outcomes, including subsequent patterns of recommended care delivery, remain underexplored. To improve outcomes among high-risk subgroups interfacing with radiation oncology, including older adults with NSCLC undergoing SBRT, further interrogation of these practical factors is needed.

Finally, the investigators will use facial photographs and audio-visual data from the PGA to develop and evaluate artificial intelligence algorithm(s) to identify vulnerable patients who might benefit from additional supportive care services.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old at time of study enrollment.
* Radiographically or pathologically confirmed stage I-II non-small cell lung cancer.
* All patients must have undergone appropriate complete imaging of their cancer consistent with the standard of care.
* Patient is expected to undergo stereotactic body radiation therapy (SBRT)
* Able to read questions in English or willing to complete survey questionnaires with the assistance of an interpreter.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Rate of referral to recommended supportive care services | One-month post PGA Implementation
  The primary endpoint for this study will be rate of referral to recommended supportive care services as compared to reported rates in historical cohorts, one month after PGA intervention.

SECONDARY OUTCOMES:
Patient acceptance of PGA usage | One-month post PGA Implementation
  The secondary endpoint for this study will be patient acceptance of PGA usage, as quantified by scores on the Response Burden Questionnaire (RBQ).
  Response Burden Questionnaire (RBQ)
  1. How well did these questions relate to your actual concerns?
     a. 0 (not at all related) to 10 (very related)
  2. How well did these questions describe your health and well-being?
     a. 0 (not at all related) to 10 (very related)
  3. How comfortable were you in answering these questions?
     a. 0 (not at all related) to 10 (very related)
  4. How did you feel about the length of time to complete these questions?
     a. 1 (much too long), 2 (a bit too long), 3 (just right/no problem)
  5. What questions seemed unimportant or repetitive: ______________
  6. What additional information should we gather? __________________

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No